CLINICAL TRIAL: NCT02524626
Title: Anti-inflammatory Effect of Peroperative Stimulation of the Vagus Nerve: A Potential New Therapeutical Intervention for Shortening Postoperative Ileus
Brief Title: Anti-inflammatory Effect of Peroperative Stimulation of the Vagus Nerve
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S56309
Record Dates: First submitted 2015-05-07; First posted 2015-08-17 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Ileus
Keywords: Vagus nerve stimulation; Postoperative ileus
MeSH Terms: interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham stimulation (Sham Comparator): no stimulation of vagus nerve
  Interventions: Procedure: Sham stimulation
- Vagus stimulation (Active Comparator): Stimulation of the vagus nerve at the beginning and the end of the surgery
  Interventions: Procedure: Vagus stimulation

INTERVENTIONS:
Procedure: Sham stimulation — Sham stimulation
  Arms: Sham stimulation
Procedure: Vagus stimulation — Vagus stimulation
  Arms: Vagus stimulation

SUMMARY:
Hypothesis:

Electrical stimulation of the abdominal vagus nerve has anti-inflammatory effects which lead to a faster postoperative recovery after abdominal surgery.

Aims:

In the present study, the investigators want evaluate the anti-inflammatory effect of peroperative electrical stimulation of the vagus nerve. In addition, the investigators want to determine whether vagus nerve stimulation leads to a faster postoperative recovery. To this end, the following aims are formulated:

1. to determine whether vagus nerve stimulation leads to an improvement in gastrointestinal transit using radiological testing
2. to evaluate whether electrical stimulation of the vagus nerve leads to clinical improvement (daily questionnaire)
3. to show that electrical stimulation of the intra-abdominal vagus nerve reduces the inflammatory response to abdominal surgery

ELIGIBILITY:
Inclusion Criteria:

* patients with ovarium, pancreas or colorectal carcinoma eligible for resection

Exclusion Criteria:

* preoperative therapeutic abdominal radiation shorter than 2 weeks prior to surgery
* evident intra-abdominal inflammation (diagnosed by imaging and/or laboratory test results, including abscess or cholecystitis)
* American Society of Anesthesiologists physical-health status classification (ASA-PS) > 3
* poorly regulated diabetes (> 200 mg/dl (= 11 mmol/l)
* surgery due to chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The gastrointestinal transit (geometric mean) | From postoperative day 3 until postoperative day 7

SECONDARY OUTCOMES:
Gastric stasis (volume of gastric fluid produced by gastric tube on postoperative day 1 | From the date of surgery until postoperative day 1
Time to first flatus | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to tolerance of oral food intake | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to tolerance of oral food intake and first defecation | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to first defecation | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Gastrointestinal symptoms (nausea, pain, vomiting, bloating) | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to discharge from the hospital | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Levels of pro-inflammatory cytokines in intestinal tissue, serum, peritoneal lavage and supernatant of stimulated whole blood | From the date of surgery until the date of lab analysis (up to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, M.D., Principal Investigator — Catholic University Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Kalff JC, Buchholz BM, Eskandari MK, Hierholzer C, Schraut WH, Simmons RL, Bauer AJ. Biphasic response to gut manipulation and temporal correlation of cellular infiltrates and muscle dysfunction in rat. Surgery. 1999 Sep;126(3):498-509. PMID 10486602
- [Background] Kalff JC, Schraut WH, Simmons RL, Bauer AJ. Surgical manipulation of the gut elicits an intestinal muscularis inflammatory response resulting in postsurgical ileus. Ann Surg. 1998 Nov;228(5):652-63. doi: 10.1097/00000658-199811000-00004. PMID 9833803